CLINICAL TRIAL: NCT02731404
Title: The Effects of High Frequency Jet Ventilation on Intra-ocular Pressure During Laparoscopic Operations (Lap. Cholecystectomy) With Positive Pressure Pneumoperitoneum
Brief Title: Intra-ocular Pressure and Ventilation
Acronym: pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Amitai Bickel MD, Primary Investigator, Western Galilee Hospital-Nahariya
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: NHR-12-0094
Record Dates: First submitted 2016-03-22; First posted 2016-04-07 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Pneumoperitoneum
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IPPV ventilation (Other): standard intermittent positive pressure ventilation in patients undergoing laparoscopic cholecystectomy
  Interventions: Procedure: IPPV ventilation
- HFJV ventilation (Other): high frequency jet ventilation in patients undergoing laparoscopic cholecystectomy
  Interventions: Procedure: HFJV ventilation

INTERVENTIONS:
Procedure: HFJV ventilation — The investigators used the Perkins tonometer for monitoring intra-ocular pressure. Evaluation of intra-ocular pressure was done before induction of anesthesia, end of induction, during surgery and at the end of surgery.
  Arms: HFJV ventilation
Procedure: IPPV ventilation — The investigators used the Perkins tonometer for monitoring intra-ocular pressure. Evaluation of intra-ocular pressure was done before induction of anesthesia, end of induction, during surgery and at the end of surgery.
  Arms: IPPV ventilation

SUMMARY:
Background: Positive pressure pneumoperitoneum (PP) may involve adverse pathophysiological changes, including increased intra-thoracic and ocular pressure, when combined with standard ventilation. High frequency jet ventilation (HFJV) was reported to reduce the adverse cardiovascular effects during laparoscopic cholecystectomy.

Aim: To study the effects of HFJV on intra-ocular pressure changes (reflecting intra-cranial pressure) during laparoscopic surgery under PP.

DETAILED DESCRIPTION:
Patients and methods: The investigators studied 2 groups of patients electively scheduled for laparoscopic cholecystectomy. The study group included 10 patients that were ventilated by high frequency jet ventilation (HFJV). In the control group (16 patients) the investigators used the standard intermittent positive pressure ventilation (IPPV). Both groups were matched according to clinical and hemodynamic parameters. Intra-ocular pressure was measured by a senior ophthalmologist that was blinded to the ventilation technique. Laparoscopic surgery was done as usual, and the intra-peritoneal pressure was automatically set on 14 mmHg. Statistical significance was considered whenever P value was less than 0.05.

The investigators anticipate that the use of HFJV during laparoscopic operations under PP may prevent increased intra-ocular pressure that accompanies increased intra-abdominal pressure under conventional ventilation (IPPV).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective laparoscopic cholecystectomy

Exclusion Criteria:

* Ophthalmologic and severe Cardiopulmonary diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Intra-ocular pressure | During procedure

CONTACTS AND LOCATIONS:
Overall Officials: Amitai Bickel, MD, Principal Investigator — Western Galilee Hospital, Bar Ilan Faculty of Medicine